CLINICAL TRIAL: NCT06066567
Title: INFLUENCE of COMBINED INTERFERENTIAL CURRENT STIMULATION and ABDOMINAL DRAW-IN EXERCISES in the TREATMENT of CHRONIC NON-SPECIFIC LOW BACK PAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Rafat, Lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004618
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: To Investigate Influence of a Combined Interferential Current Stimulation and Abdominal Draw -in Exercises in Patients with Chronic N
MeSH Terms: interventions — Electric Stimulation Therapy; Exercise Therapy; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: treatment group (Experimental)
  Interventions: Device: Interferential current stimulation; Other: Draw- In exercises,,
- control group (Active Comparator)
  Interventions: Other: Draw- In exercises,,

INTERVENTIONS:
Device: Interferential current stimulation — IF Current parameters will be applied as follow: Amplitude modulated frequency (AMF) 30Hz, Autosweep-5 sec, Dose-15 minutes, type of current dynamic vector field (Mitra, 2006), three days per week over four weeks (Corrêa et al., 2016) and current intensity will be increased gradually, according to the subject's condition
  Other Names: Draw- In exercises,,; hot pack; back muscles stretching; strengthening exercises for the back and abdominal muscles.
  Arms: Experimental: treatment group
Other: Draw- In exercises,, — From prone position, participants will lay face down on the bed and flexed their hips and knees at 0°. A PBU will be positioned below the pubis symphysis with the decreasing edge consistent with the ASIS and will be overstated to 70 mmHg. The participants will be trained to gently draw in the lower part of the abdomen under the navel. In addition, while maintaining the neutral pelvic position, the movement of the upper part of the abdomen will be restricted so that the pressure will be decreased by approximately 10 mmHg. The participants will maintain this position for 10 s
  Other Names: back muscles stretching; strengthening exercises for the back and abdominal muscles.; hot pack

SUMMARY:
The purpose of this study is to investigate influence of a combined interferential (IF) current stimulation and abdominal draw-in exercises on the abdominal muscle thickness, TrA endurance, pain intensity and function disability in patients with chronic non-specific LBP (CNSLBP) CNSLBP is considered the second most common health problem after headache. The lifetime of LBP among Egyptian patients in a family center reached 48%, which indicates that LBP is a prevalent symptom that deserves more attention.

One hypothesis for the development of LBP is due to a dysfunction in the control of the abdominal and back muscles and this change in spinal control is due in part to in local segmental muscles dysfunction, such as the transversus abdominis (TrA). Interferential therapy (IFT) is capable of achieving uniform stimulation and high reproducibility, it is thought to be less stressful, as well as enhance deep muscle contraction.

Also, there is the specific training of the TrA provided functional and therapeutic benefits, such as unloading of the spine, anticipatory postural control, intersegmental stabilization of the spine, and long-term pain relief. Draw-in is a typical TrA exercise.

Many studies have mainly focused on the morphological aspects of paraspinal muscles which play an essential role in patients with CNSLBP while our study focused on influence of a combined IFT stimulation and abdominal draw-in exercises on the abdominal muscle thickness, TrA endurance, pain intensity and function disability in patients with chronic non-specific LBP (CNSLBP

DETAILED DESCRIPTION:
60 patients suffering from chronic non-specific low back pain will participate in this study. Both sexes will participate in this study; aged 20-45 years. will be diagnosed and referred from Orthopedist. The study will be conducted at outpatient clinic of Deraya university Elmina government. The patients will be divided randomly into two groups equal in numbers (group A), (group B).

Group(A): (Experimental group) :( 30 patients will receive IFC stimulation, Draw In exercises from prone position, hot pack, back muscles stretching and strengthening exercises for the back and abdominal muscles).

Group(B): (control group) (30 patients will receive Draw In exercises from prone position, hot pack, back muscles stretching and strengthening exercises for the back and abdominal muscles).

ELIGIBILITY:
Inclusion Criteria:

* 60 patients with chronic non-specific low back pain (>3 months).
* 2. Age of participants will range from 20 to 45 years.
* 3.Both sexes will participate in this study.
* 4.Body mass index (BMI) will range from 25 to 29.9 (Kg / m2).

Exclusion Criteria:

* Subjects will be excluded from the study if they have previous spinal surgery, spinal cord injury or unstable neurological signs, Lumbar intervertebral disc, congenital postural deformities, inability to contract the abdominal muscles, cauda equine symptoms related to the spine including changes in bowel and bladder control, cardiac pacemaker, and females during pregnancy.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Abdominal muscle thickness | 4 weeks
  TrA, External Oblique (EO) and Internal Oblique (IO) with Ultrasonography imaging examination.
Transverse abdominis (TrA) muscle endurance | 4 weeks
  Transverse abdominis (TrA) muscle endurance with prone endurance test guided by Pressure Biofeedback Unit (PBU).
Pain intensity | 4 weeks
  Pain intensity with visual analogue scale (VAS).
. Functional disability | 4 weeks
  Functional disability with Arabic version of Oswestry Disability Index (ODI).

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Cairo University, Giza, Giza Governorate
  - Faculty of physical therapy, Giza

IPD SHARING:
Plan to Share IPD: No